CLINICAL TRIAL: NCT01214265
Title: A Pilot Clinical Study to Evaluate the Initial Feasibility of Neuromodulation Therapy in Treating Patients With Overactive Bladder Via Magnetic Stimulation of the Posterior Tibial Nerve
Brief Title: A Clinical Study for Magnetic Stimulation of the Posterior Tibial Nerve in Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EMKinetics, Inc (Industry)
Responsible Party: Amit Rajguru, MD, EMKinetics, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMK0708C
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EMKinetics non-invasive Magnetic neurostimulator — Patients will be treated with 12 weekly sessions of magnetic stimulation of the posterior tibial nerve at 20 hz using the EMKinetics non-invasive Magnetic neurostimulator.

SUMMARY:
To evaluate the safety and feasibility of non-invasive magnetic stimulation of the posterior tibial nerve using the EMKinetics LoFIT Pulse System for treating patients with documented overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age
* A score of > 4 on the OAB-q short form for urgency (question 1)
* Average urinary frequency > 10 times in one 24 hour day based on a 3-day voiding diary
* Self-reported bladder symptoms present > 3 months
* Self-reported failed conservative care (e.g., dietary restriction, fluid restriction, bladder training, behavioral modification, pelvic muscle training, biofeedback, etc.) or use of antimuscarinics.
* Off all anti-muscarinics for at least 2 weeks prior to enrollment
* Capable of giving informed consent
* Ambulatory and able to use a toilet independently, without difficulty
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* The patient is pregnant or intends to become pregnant during the course of the study. (Patients becoming pregnant during the course of the study will immediately be terminated from the study.)
* The patient has an active urinary tract infection.
* Neurogenic bladder
* Botox use in bladder or pelvic floor muscles in the past year
* Pacemakers or implantable defibrillators
* Primary complaint of stress urinary incontinence
* Current vaginal infection
* Current use of InterStim
* Current use of Bion
* Current use of TENS in the pelvic region, back or leg
* Previously been treated with PTNS
* Use of investigational drug/device therapy within the past 4 weeks
* Participating or have participated within the past 4 weeks in any clinical investigation involving or impacting gynecologic, urinary or renal function
* Deemed unsuitable for enrollment in study by the investigators based on subjects' history or physical examination
* The patient has metal implant from surgery or a metallic foreign body in either leg below (distal to) the knee (or permanent metallic tattoo <30cm from left ankle).
* The patient has chronic constipation (less than two (2) bowel movements per week)
* The patient has history of gastric or urinary retention
* The patient has uncontrolled diabetes
* Subjects with nerve damage, injury or surgery that would impact either tibial nerve or pelvic floor function
* The patient is unable or unwilling to sign informed consent
* The patient is currently on pharmacologic treatment that could affect bladder function
* Known Cystocele >/= to Grade 3 that has not been reduced by treatment (surgery or pessary)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Global Response Assessment | After 12 weeks of therapy
  Improved score on the Global Response Assessment (GRA) scale after 12 weeks of therapy. A score of 2 (moderately improved) or 3 (markedly improved) constitutes a responder on the 7 point scale

SECONDARY OUTCOMES:
Urinary Frequency | After 12 weeks of therapy
  Change in Urinary Frequency (Voiding Diary) from Baseline to 12 weeks
Urinary Incontinence | After 12 weeks of therapy
  Change in Urinary Incontinence (Voiding Diary) from Baseline to 12 weeks
Overactive Bladder Symptoms (OAB-q SF) | After 12 weeks of therapy
  Change in Overactive Bladder Symptoms (OAB-q SF) from Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Incontinence and Pelvic Support Institute, Mission Viejo, California, United States